CLINICAL TRIAL: NCT02416037
Title: Trans-Pulmonary Pressure and Prone Position in Ards Patients
Brief Title: Trans-pulmonary Pressure in ARDS
Acronym: T3P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL14-0333
Record Dates: First submitted 2015-04-03; First posted 2015-04-14 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; prone position; PEEP; mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prone Proseva (Experimental)
  Interventions: Device: level of positive end expiratory pressure (Prone Proseva)
- Prone Talmor (Active Comparator)
  Interventions: Device: level of positive end expiratory pressure (Prone Talmor)

INTERVENTIONS:
Device: level of positive end expiratory pressure (Prone Proseva) — PEEP based on PEEP/FIO2 table vs PEEP based on the value of oesophageal pressure
  Arms: Prone Proseva
Device: level of positive end expiratory pressure (Prone Talmor) — PEEP based on PEEP/FIO2 table vs PEEP based on the value of oesophageal pressure
  Arms: Prone Talmor

SUMMARY:
Adequate PEEP selection in ARDS is still a matter of research. The main objectives of using PEEP in ARDS are improvement in oxygenation, lung recruitment at the end of expiration, prevention of opening and closing of terminal respiratory units at minimal hemodynamic compromise. The challenge is to carry out these objectives in a patient-centered approach based on individual characteristic of lung pathophysiology. Recently, it has been proposed to set PEEP from the trans-pulmonary end-expiratory pressure. Trans-pulmonary pressure (Ptp) is obtained from the difference between airway pressure and measured esophageal pressure (Pes). Measured Pes values have been found positive in the supine position in ARDS patients, leading to negative values of Ptp. The strategy proposed by Talmor and coworkers is to adjust PEEP up to get Ptp between 0 and 10 cm H2O. Whether this strategy improves survival is under investigation. Prone position ventilation significantly improves survival in severe ARDS as demonstrated by meta-analyses and a recent multicenter randomized controlled trial.

The purpose of present project is to investigate Ptp at end-expiration in the prone position in severe ARDS. The project is centered on the question about what are the values of measured Pes in prone position. The hypothesis is that they are lower than in the supine position due to the relief of the weight of heart, mediastinum and lung and also to recruitment of dorsal lung regions. To investigate this hypothesis, measured Pes, Ptp, end-expiratory lung volume, overall lung recruitment (pressure-volume curve), and regional recruitment by using electrical impedance tomography. will be assessed in supine then in the prone position across two different strategies of PEEP selection, PEEP/FIO2 table and Talmor proposal.

ELIGIBILITY:
Inclusion Criteria:

* ARDS
* intubated
* indication of proning
* no contra-indication of proning

Exclusion Criteria:

* contra-indication to proning
* contra-indication to esophageal balloon
* proning before
* end of life decision
* legal protection
* pregnancy
* ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Value of the esophageal pressure measured at the end of expiration | 6.5 hours after inclusion
  Oesophageal pressure is measured from a balloon inserted into the mid oesophagus at the end of expiration. Its value is subtracted to the airway pressure at the end of expiration leading to trans-pulmonary pressure at the end of expiration (Ptp,ee). The measurements are done first in the supine position. In the standardized condition PEEP is set from a PEEP/FIO2 table and Ptp,ee is measured. In the Talmor approach PEEP is set to obtain Ptp,ee between 0 and 10 cm H2O. The patient is then turned to the prone position. The measurements are repeated in the same way. Then for the rest of the proning session the patient receive either level of PEEP from each strategy. Measurements are repeated at the end of the session.
Value of the esophageal pressure measured at the end of expiration | 8.0 hours after inclusion
  Oesophageal pressure is measured from a balloon inserted into the mid oesophagus at the end of expiration. Its value is subtracted to the airway pressure at the end of expiration leading to trans-pulmonary pressure at the end of expiration (Ptp,ee). The measurements are done first in the supine position. In the standardized condition PEEP is set from a PEEP/FIO2 table and Ptp,ee is measured. In the Talmor approach PEEP is set to obtain Ptp,ee between 0 and 10 cm H2O. The patient is then turned to the prone position. The measurements are repeated in the same way. Then for the rest of the proning session the patient receive either level of PEEP from each strategy. Measurements are repeated at the end of the session.
Value of the esophageal pressure measured at the end of expiration | 10 hours after inclusion
  Oesophageal pressure is measured from a balloon inserted into the mid oesophagus at the end of expiration. Its value is subtracted to the airway pressure at the end of expiration leading to trans-pulmonary pressure at the end of expiration (Ptp,ee). The measurements are done first in the supine position. In the standardized condition PEEP is set from a PEEP/FIO2 table and Ptp,ee is measured. In the Talmor approach PEEP is set to obtain Ptp,ee between 0 and 10 cm H2O. The patient is then turned to the prone position. The measurements are repeated in the same way. Then for the rest of the proning session the patient receive either level of PEEP from each strategy. Measurements are repeated at the end of the session.
Value of the esophageal pressure measured at the end of expiration | 11.5 hours after inclusion
  Oesophageal pressure is measured from a balloon inserted into the mid oesophagus at the end of expiration. Its value is subtracted to the airway pressure at the end of expiration leading to trans-pulmonary pressure at the end of expiration (Ptp,ee). The measurements are done first in the supine position. In the standardized condition PEEP is set from a PEEP/FIO2 table and Ptp,ee is measured. In the Talmor approach PEEP is set to obtain Ptp,ee between 0 and 10 cm H2O. The patient is then turned to the prone position. The measurements are repeated in the same way. Then for the rest of the proning session the patient receive either level of PEEP from each strategy. Measurements are repeated at the end of the session.
Value of the esophageal pressure measured at the end of expiration | up to 26.5 hours after inclusion
  Oesophageal pressure is measured from a balloon inserted into the mid oesophagus at the end of expiration. Its value is subtracted to the airway pressure at the end of expiration leading to trans-pulmonary pressure at the end of expiration (Ptp,ee). The measurements are done first in the supine position. In the standardized condition PEEP is set from a PEEP/FIO2 table and Ptp,ee is measured. In the Talmor approach PEEP is set to obtain Ptp,ee between 0 and 10 cm H2O. The patient is then turned to the prone position. The measurements are repeated in the same way. Then for the rest of the proning session the patient receive either level of PEEP from each strategy. Measurements are repeated at the end of the session.

SECONDARY OUTCOMES:
Elastance of the chest wall | 6.5 hours after inclusion
  The elastance of the chest wall is the change in esophageal pressure between expiration and inspiration in response to a change in lung volume. It is not substantially changed by PEEP but it is by the change in position.
Elastance of the chest wall | 8.0 hours after inclusion
  The elastance of the chest wall is the change in esophageal pressure between expiration and inspiration in response to a change in lung volume. It is not substantially changed by PEEP but it is by the change in position.
Elastance of the chest wall | 10 hours after inclusion
  The elastance of the chest wall is the change in esophageal pressure between expiration and inspiration in response to a change in lung volume. It is not substantially changed by PEEP but it is by the change in position.
Elastance of the chest wall | 11.5 hours after inclusion
  The elastance of the chest wall is the change in esophageal pressure between expiration and inspiration in response to a change in lung volume. It is not substantially changed by PEEP but it is by the change in position.
Elastance of the chest wall | up to 26.5 hours after inclusion
  The elastance of the chest wall is the change in esophageal pressure between expiration and inspiration in response to a change in lung volume. It is not substantially changed by PEEP but it is by the change in position.
Transpulmonary pressure at the end of expiration (Ptp,ee) | 6.5 hours after inclusion
  In the standardized condition, either in supine or prone, the transpulmonary pressure is the difference between airway pressure and esophageal pressure at the end of expiration. In the standardized approach, PEEP is set according to a PEEP/FIO2 table and Ptp,ee is dependent on the PEEP/FIO2 table. With the Talmor approach, Ptp,ee is directly set from measurement of esophageal pressure and PEEP set according to the PEEP/FIO2 table.
Transpulmonary pressure at the end of expiration (Ptp,ee) | 8.0 hours after inclusion
  In the standardized condition, either in supine or prone, the transpulmonary pressure is the difference between airway pressure and esophageal pressure at the end of expiration. In the standardized approach, PEEP is set according to a PEEP/FIO2 table and Ptp,ee is dependent on the PEEP/FIO2 table. With the Talmor approach, Ptp,ee is directly set from measurement of esophageal pressure and PEEP set according to the PEEP/FIO2 table.
Transpulmonary pressure at the end of expiration (Ptp,ee) | 10 hours after inclusion
  In the standardized condition, either in supine or prone, the transpulmonary pressure is the difference between airway pressure and esophageal pressure at the end of expiration. In the standardized approach, PEEP is set according to a PEEP/FIO2 table and Ptp,ee is dependent on the PEEP/FIO2 table. With the Talmor approach, Ptp,ee is directly set from measurement of esophageal pressure and PEEP set according to the PEEP/FIO2 table.
Transpulmonary pressure at the end of expiration (Ptp,ee) | 11.5 hours after inclusion
  In the standardized condition, either in supine or prone, the transpulmonary pressure is the difference between airway pressure and esophageal pressure at the end of expiration. In the standardized approach, PEEP is set according to a PEEP/FIO2 table and Ptp,ee is dependent on the PEEP/FIO2 table. With the Talmor approach, Ptp,ee is directly set from measurement of esophageal pressure and PEEP set according to the PEEP/FIO2 table.
Transpulmonary pressure at the end of expiration (Ptp,ee) | up to 26.5 hours after inclusion
  In the standardized condition, either in supine or prone, the transpulmonary pressure is the difference between airway pressure and esophageal pressure at the end of expiration. In the standardized approach, PEEP is set according to a PEEP/FIO2 table and Ptp,ee is dependent on the PEEP/FIO2 table. With the Talmor approach, Ptp,ee is directly set from measurement of esophageal pressure and PEEP set according to the PEEP/FIO2 table.
End expiratory lung volume (EELV) | 6.5 hours after inclusion
  EELV is the volume of gas at the end of expiration. It is measured from the ventilator by using the washout-washin technique after a small change in the FIO2. An increase in EELV can indicate recruitment (reopening of non aerated lung tissue) but some overinflation may also contribute to this increase. PEEP and prone position can increase EELV.
End expiratory lung volume (EELV) | 8.0 hours after inclusion
  EELV is the volume of gas at the end of expiration. It is measured from the ventilator by using the washout-washin technique after a small change in the FIO2. An increase in EELV can indicate recruitment (reopening of non aerated lung tissue) but some overinflation may also contribute to this increase. PEEP and prone position can increase EELV.
End expiratory lung volume (EELV) | 10 hours after inclusion
  EELV is the volume of gas at the end of expiration. It is measured from the ventilator by using the washout-washin technique after a small change in the FIO2. An increase in EELV can indicate recruitment (reopening of non aerated lung tissue) but some overinflation may also contribute to this increase. PEEP and prone position can increase EELV.
End expiratory lung volume (EELV) | 11.5 hours after inclusion
  EELV is the volume of gas at the end of expiration. It is measured from the ventilator by using the washout-washin technique after a small change in the FIO2. An increase in EELV can indicate recruitment (reopening of non aerated lung tissue) but some overinflation may also contribute to this increase. PEEP and prone position can increase EELV.
End expiratory lung volume (EELV) | up to 26.5 hours after inclusion
  EELV is the volume of gas at the end of expiration. It is measured from the ventilator by using the washout-washin technique after a small change in the FIO2. An increase in EELV can indicate recruitment (reopening of non aerated lung tissue) but some overinflation may also contribute to this increase. PEEP and prone position can increase EELV.
Regional lung ventilation | 6.5 hours after inclusion
  regional ventilation is measured by using electrical impedance tomography. The change in thoracic impedance in response to electric current of small amplitude (50 ms) is proportional to amount of air among other factors, which are less important in magnitude as compared to air. The lung is sampled into anterior and posterior regions. The location of better aeration with PEEP and position will be mapped.
Regional lung ventilation | 8.0 hours after inclusion
  regional ventilation is measured by using electrical impedance tomography. The change in thoracic impedance in response to electric current of small amplitude (50 ms) is proportional to amount of air among other factors, which are less important in magnitude as compared to air. The lung is sampled into anterior and posterior regions. The location of better aeration with PEEP and position will be mapped.
Regional lung ventilation | 10 hours after inclusion
  regional ventilation is measured by using electrical impedance tomography. The change in thoracic impedance in response to electric current of small amplitude (50 ms) is proportional to amount of air among other factors, which are less important in magnitude as compared to air. The lung is sampled into anterior and posterior regions. The location of better aeration with PEEP and position will be mapped.
Regional lung ventilation | 11.5 hours after inclusion
  regional ventilation is measured by using electrical impedance tomography. The change in thoracic impedance in response to electric current of small amplitude (50 ms) is proportional to amount of air among other factors, which are less important in magnitude as compared to air. The lung is sampled into anterior and posterior regions. The location of better aeration with PEEP and position will be mapped.
Regional lung ventilation | up to 26.5 hours after inclusion
  regional ventilation is measured by using electrical impedance tomography. The change in thoracic impedance in response to electric current of small amplitude (50 ms) is proportional to amount of air among other factors, which are less important in magnitude as compared to air. The lung is sampled into anterior and posterior regions. The location of better aeration with PEEP and position will be mapped.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital de la Croix-Rousse, Lyon

REFERENCES:
- [Result] Mezidi M, Parrilla FJ, Yonis H, Riad Z, Bohm SH, Waldmann AD, Richard JC, Lissonde F, Tapponnier R, Baboi L, Mancebo J, Guerin C. Effects of positive end-expiratory pressure strategy in supine and prone position on lung and chest wall mechanics in acute respiratory distress syndrome. Ann Intensive Care. 2018 Sep 10;8(1):86. doi: 10.1186/s13613-018-0434-2. PMID 30203117